CLINICAL TRIAL: NCT06104982
Title: The Effect of Superimposed Electrical Stimulation on Sitting Balance, Respiratory Functions, and Abdominal Muscle Thickness in Complete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Handan Elif Nur BAYRAKTAR, Specialist Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-DRHENY-01
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injury Thoracic
Keywords: spinal cord injury; abdominal muscle; electrical stimulation; sitting balance
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Investigators included thirty-four participants with thoracic complete SCI in this randomized controlled and prospective study. Investigators divided the participants into two equal groups, where one group received the biofeedback triggered superimposed functional electrical stimulation (SiFES) applied to the abdominal muscles, and the control group received transcutaneous electrical stimulation (TE) only, applied three times a week for four weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SiFES group (Experimental): The investigators applied FES to the abdominal muscles of the SiFES group bilaterally, using 2 units of NeuroTrac MyoPlus Pro single-channel electromyography biofeedback electrotherapy devices. The investigators conducted electrical stimulation for a total of 10 minutes per session, with 5 minutes dedicated to bilateral rectus abdominis (RA) and 5 minutes to bilateral obliques externus (OE), obliques internus (OI), and transversus abdominis (TA) muscles three days a week, a period of four weeks. The investigators triggered the initial contraction of the abdominal muscles by instructing the patient to slightly flex their head before the application of electrical stimulation. During this process, the contraction was detected by the surface EMG present in the FES device, and the abdominal muscles were stimulated with electrical impulses.
  Interventions: Device: NeuroTrac MyoPlus Pro single-channel electromyography biofeedback electrotherapy devices
- Control group (TE group) (Active Comparator): The investigators administered isometric strengthening to the TE groups, three days a week, with three sets per session, a period of four weeks.
  Interventions: Other: Isometric strengthening exercises

INTERVENTIONS:
Device: NeuroTrac MyoPlus Pro single-channel electromyography biofeedback electrotherapy devices — Neuromuscular electrical stimulation (NMES) is applied to intact second motor neurons and target muscles of patients with SCI and provides functional and therapeutic benefits in neurological rehabilitation. Functional electrical stimulation (FES) is a type of NMES that is used for electrical stimulation during exercises such as crunches. Newly used SiFES is a method in which the biofeedback-enabled FES device detects muscle contractions, and this electromyography (EMG) signal triggers the muscle stimulant mode of the device.
  Arms: SiFES group
Other: Isometric strengthening exercises — Isometric abdominal strengthening exercises are part of the standard rehabilitation program for individuals with spinal cord injuries.
  Arms: Control group (TE group)

SUMMARY:
The primary aim of the current study was to investigate the effects of SiFES (superimposed functional electrical stimulation) on sitting balance in patients with complete Spinal Cord Injury (SCI) compared to exercise alone. Additionally, the study aims to investigate improvements in respiratory functions and changes in abdominal muscle thickness measured by ultrasonography (USG) following SiFES treatment.

The fundamental questions that investigators want to answer are as follows:

* [question 1]: "Does abdominal SiFES therapy improve sitting balance in patients with complete SCI?"
* [question 2]: "Does abdominal SiFES therapy improve respiratory functions in patients with complete SCI?"

DETAILED DESCRIPTION:
Many patients with SCI are ambulatory with a wheelchair. Therefore, providing good sitting balance in these patients is a key factor for performing activities of daily living (ADL) and achieving functional independence. Paralysis of abdominal muscles in patients with SCI disrupts body balance. In these patients, problems with trunk balance can lead to frequent falls and poor rehabilitation outcomes. Also, abdominal muscles assist in forceful expiration. Loss of innervation to abdominal and intercostal muscles reduces their ability to excrete secretions and cough effectively. As a result, respiratory tract complications, such as pneumonia, atelectasis, and respiratory failure can arise. It should be noted that in individuals with SCI, respiratory tract complications are the primary cause of morbidity and mortality. Newly used SiFES is a method in which the biofeedback-enabled FES device detects muscle contractions, and this electromyography (EMG) signal triggers the muscle stimulant mode of the device. In this method, more stimuli are conveyed to the brain through afferent nerves, allowing for motor learning to potentially occur by reviving the region represented in the cortex. In the current study, the investigators planned due to the anticipation that the synchronized stimulation of SiFES with function will be effective in patients with SCI injuries who currently have weak contraction abilities. The investigators considering the key role of abdominal muscles in trunk stability, believed that the integrated effect of SiFES is of great importance to patients. In the current randomized controlled and prospective study, the investigators included thirty-four participants with thoracic complete SCI. The investigators divided the participants into two equal groups: one group received SiFES applied to the abdominal muscles, while the control group received therapeutic exercise (TE) only. The investigators administered the interventions three times a week for four weeks. The investigators conducted muscle thickness measurements of bilateral rectus abdominis (RA), obliques externus (OE), obliques internus (OI), and transversus abdominis (TA) muscles using ultrasonography for all participants before and after treatment. Additionally, the investigators applied the modified functional reach test (mFRT), trunk control test (TCT), and pulmonary function test (PFT) to assess the participants.

ELIGIBILITY:
Inclusion Criteria:

* being between 18-65 years old
* having a minimum of 3 months since the spinal cord injury
* having complete paraplegia according American Spinal Injury Association (ASIA) disorder scale A due to traumatic spinal cord injury
* being able to sit unsupported in a wheelchair

Exclusion Criteria:

* malignancy,
* epilepsy, heart failure,
* intracardiac defibrillator (ICD)
* an open wound in the application area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-06 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Modified Functional Reach Test (mFRT) (reaching of forward, right, left) | Baseline - week 4
  The mFRT, which is a validated and reliable tool for measuring sitting balance in patients with SCI was used in this study. Before the investigators conducted the test, the participant was positioned in an upright sitting posture in a wheelchair. The investigators took measurements in three directions: forward reach (using the dominant extremity), right reach, and left reach, both before and after the treatment, for both groups. During the modified functional reach test, the participants reached out as far as possible in the forward, right, and left directions. The investigators repeated the test three times, and there was a 5-minute interval between each repetition. The investigators recorded the best measurement out of the three trials in centimeters.

SECONDARY OUTCOMES:
Abdominal muscle thickness, the thicknesses of the right and left rectus abdominis (RA), obliques externus (OE), obliques internus (OI), and transversus abdominis (TA) | Baseline - week 4
  The investigators conducted muscle thickness measurements using an 8-12 megahertz (MHz) linear probe on a real-time B mode USG device (GE LOGIQ 7, General Electric Co., Wisconsin, USA). The investigators took measurements at the end of expiration while the patient was lying on their back, with their body exposed and a pillow placed under their head. The investigators applied gel between the probe and the skin to ensure proper contact and accurate measurements. To measure the RA thickness, two centimeters lateral to the umbilicus were marked on both the right and left sides. To measure the thicknesses of the OE, OI, and TA muscles, the lowest point of the 11th rib and the midpoint of the iliac crest were marked on both the right and left sides at the level of the anterior axillary line. The investigators took three measurements from these marked points both before and after the treatment, and recorded the average of these measurements in centimeters.
Trunk Control Test (TCT), | Baseline - week 4
  The TCT is a test with proven validity and reliability, used to measure trunk balance in patients with SCI. The investigators conducted TCT both before and after the treatment in both groups. The TCT comprises two parts: static and dynamic balance assessments, which involve reaching for variable targets and assuming required positions. The investigators evaluated participants using a scoring system ranging from 0 to 24, both before and after the treatment. The score reflects their performance in maintaining trunk balance, with higher scores indicating better trunk control.
Forced expiratory volume in one second (FEV1) | Baseline - week 4
  The PFT is a laboratory method used for diagnosing and monitoring lung diseases, and objectively evaluating lung functions. In the current study, the investigators measured the PFT by the same person before and after treatment in both groups, using a simple spirometer device (COSMED, Pony FX) at the Ankara City Hospital Physical Therapy Hospital Cardiopulmonary Rehabilitation Unit. The investigators conducted the PFT three times for each participant and recorded the best spirogram image. From these spirometry results, the investigators recorded the FEV1.
Forced vital capacity (FVC) | Baseline - week 4
  The PFT is a laboratory method used for diagnosing and monitoring lung diseases, and objectively evaluating lung functions. In the current study, the investigators measured the PFT by the same person before and after treatment in both groups, using a simple spirometer device (COSMED, Pony FX) at the Ankara City Hospital Physical Therapy Hospital Cardiopulmonary Rehabilitation Unit. The investigators conducted the PFT three times for each participant and recorded the best spirogram image. From these spirometry results, the investigators recorded the FVC.
FEV1/FVC | Baseline - week 4
  The PFT is a laboratory method used for diagnosing and monitoring lung diseases, and objectively evaluating lung functions. In the current study, the investigators measured the PFT by the same person before and after treatment in both groups, using a simple spirometer device (COSMED, Pony FX) at the Ankara City Hospital Physical Therapy Hospital Cardiopulmonary Rehabilitation Unit. The investigators conducted the PFT three times for each participant and recorded the best spirogram image. From these spirometry results, the investigators recorded the FEV1/FVC.
Peak expiratory flow rate (PEF) | Baseline - week 4
  The PFT is a laboratory method used for diagnosing and monitoring lung diseases, and objectively evaluating lung functions. In the current study, the investigators measured the PFT by the same person before and after treatment in both groups, using a simple spirometer device (COSMED, Pony FX) at the Ankara City Hospital Physical Therapy Hospital Cardiopulmonary Rehabilitation Unit. The investigators conducted the PFT three times for each participant and recorded the best spirogram image. From these spirometry results, the investigators recorded the PEF.
The flow rate between 25% and 75% of FVC (PEF 25%-75%) | Baseline - week 4
  The PFT is a laboratory method used for diagnosing and monitoring lung diseases, and objectively evaluating lung functions. In the current study, the investigators measured the PFT by the same person before and after treatment in both groups, using a simple spirometer device (COSMED, Pony FX) at the Ankara City Hospital Physical Therapy Hospital Cardiopulmonary Rehabilitation Unit. The investigators conducted the PFT three times for each participant and recorded the best spirogram image. From these spirometry results, the investigators recorded the PEF 25%-75%.
Maximum voluntary ventilation (MVV) | Baseline - week 4
  The PFT is a laboratory method used for diagnosing and monitoring lung diseases, and objectively evaluating lung functions. In the current study, the investigators measured the PFT by the same person before and after treatment in both groups, using a simple spirometer device (COSMED, Pony FX) at the Ankara City Hospital Physical Therapy Hospital Cardiopulmonary Rehabilitation Unit. The investigators conducted the PFT three times for each participant and recorded the best spirogram image. From these spirometry results, the investigators recorded the MVV.
Vital capacity (VC) | Baseline - week 4
  The PFT is a laboratory method used for diagnosing and monitoring lung diseases, and objectively evaluating lung functions. In the current study, the investigators measured the PFT by the same person before and after treatment in both groups, using a simple spirometer device (COSMED, Pony FX) at the Ankara City Hospital Physical Therapy Hospital Cardiopulmonary Rehabilitation Unit. The investigators conducted the PFT three times for each participant and recorded the best spirogram image. From these spirometry results, the investigators recorded the VC.
Inspiratory capacity (IC) | Baseline - week 4
  The PFT is a laboratory method used for diagnosing and monitoring lung diseases, and objectively evaluating lung functions. In the current study, the investigators measured the PFT by the same person before and after treatment in both groups, using a simple spirometer device (COSMED, Pony FX) at the Ankara City Hospital Physical Therapy Hospital Cardiopulmonary Rehabilitation Unit. The investigators conducted the PFT three times for each participant and recorded the best spirogram image. From these spirometry results, the investigators recorded the IC.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Arsh A, Darain H, Rahman MU, Ullah I, Shakil-Ur-Rehman S. Reliability of modified functional reach test in the assessment of balance function in people with spinal cord injury: A systematic review. J Pak Med Assoc. 2021 Aug;71(8):2040-2044. doi: 10.47391/JPMA.1276. PMID 34418026
- [Background] McCaughey EJ, Borotkanics RJ, Gollee H, Folz RJ, McLachlan AJ. Abdominal functional electrical stimulation to improve respiratory function after spinal cord injury: a systematic review and meta-analysis. Spinal Cord. 2016 Sep;54(9):628-39. doi: 10.1038/sc.2016.31. Epub 2016 Apr 12. PMID 27067658
- [Background] Hascakova-Bartova R, Dinant JF, Parent A, Ventura M. Neuromuscular electrical stimulation of completely paralyzed abdominal muscles in spinal cord-injured patients: a pilot study. Spinal Cord. 2008 Jun;46(6):445-50. doi: 10.1038/sj.sc.3102166. Epub 2008 Jan 29. PMID 18227852
- [Background] Gater DR Jr, Dolbow D, Tsui B, Gorgey AS. Functional electrical stimulation therapies after spinal cord injury. NeuroRehabilitation. 2011;28(3):231-48. doi: 10.3233/NRE-2011-0652. No abstract available. PMID 21558629
- [Background] Cheng PT, Chen CL, Wang CM, Chung CY. Effect of neuromuscular electrical stimulation on cough capacity and pulmonary function in patients with acute cervical cord injury. J Rehabil Med. 2006 Jan;38(1):32-6. doi: 10.1080/16501970510043387. PMID 16548084
- [Background] McBain RA, Boswell-Ruys CL, Lee BB, Gandevia SC, Butler JE. Abdominal muscle training can enhance cough after spinal cord injury. Neurorehabil Neural Repair. 2013 Nov-Dec;27(9):834-43. doi: 10.1177/1545968313496324. Epub 2013 Jul 24. PMID 23884017
- [Background] Bersch I, Friden J. Role of Functional Electrical Stimulation in Tetraplegia Hand Surgery. Arch Phys Med Rehabil. 2016 Jun;97(6 Suppl):S154-9. doi: 10.1016/j.apmr.2016.01.035. PMID 27233590
- [Background] Chandrasekaran S, Davis J, Bersch I, Goldberg G, Gorgey AS. Electrical stimulation and denervated muscles after spinal cord injury. Neural Regen Res. 2020 Aug;15(8):1397-1407. doi: 10.4103/1673-5374.274326. PMID 31997798
- [Background] Paillard T, Noe F, Passelergue P, Dupui P. Electrical stimulation superimposed onto voluntary muscular contraction. Sports Med. 2005;35(11):951-66. doi: 10.2165/00007256-200535110-00003. PMID 16271009
- [Background] Amerijckx C, Goossens N, Pijnenburg M, Musarra F, van Leeuwen DM, Schmitz M, Janssens L. Influence of phase of respiratory cycle on ultrasound imaging of deep abdominal muscle thickness. Musculoskelet Sci Pract. 2020 Apr;46:102105. doi: 10.1016/j.msksp.2019.102105. Epub 2019 Dec 27. PMID 32217268
- [Background] Tahan N, Khademi-Kalantari K, Mohseni-Bandpei MA, Mikaili S, Baghban AA, Jaberzadeh S. Measurement of superficial and deep abdominal muscle thickness: an ultrasonography study. J Physiol Anthropol. 2016 Aug 23;35(1):17. doi: 10.1186/s40101-016-0106-6. PMID 27553830
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Lynch SM, Leahy P, Barker SP. Reliability of measurements obtained with a modified functional reach test in subjects with spinal cord injury. Phys Ther. 1998 Feb;78(2):128-33. doi: 10.1093/ptj/78.2.128. PMID 9474105
- [Background] Quinzanos J, Villa AR, Flores AA, Perez R. Proposal and validation of a clinical trunk control test in individuals with spinal cord injury. Spinal Cord. 2014 Jun;52(6):449-54. doi: 10.1038/sc.2014.34. Epub 2014 Apr 8. PMID 24710149
- [Background] Baek SO, Cho HK, Kim SY, Jones R, Cho YW, Ahn SH. Changes in deep lumbar stabilizing muscle thickness by transcutaneous neuromuscular electrical stimulation in patients with low back pain. J Back Musculoskelet Rehabil. 2017;30(1):121-127. doi: 10.3233/BMR-160723. PMID 27341642
- [Background] Hwang UJ, Jung SH, Kim HA, Kim JH, Kwon OY. Effect of Abdominal Electrical Muscle Stimulation Training With and Without Superimposed Voluntary Muscular Contraction on Lumbopelvic Control. J Sport Rehabil. 2020 Nov 1;29(8):1137-1144. doi: 10.1123/jsr.2019-0348. Epub 2020 Jan 7. PMID 31910395
- [Background] Wakahara T, Shiraogawa A. Effects of neuromuscular electrical stimulation training on muscle size in collegiate track and field athletes. PLoS One. 2019 Nov 13;14(11):e0224881. doi: 10.1371/journal.pone.0224881. eCollection 2019. PMID 31721812
- [Background] Yablon CM, Hammer MR, Morag Y, Brandon CJ, Fessell DP, Jacobson JA. US of the Peripheral Nerves of the Lower Extremity: A Landmark Approach. Radiographics. 2016 Mar-Apr;36(2):464-78. doi: 10.1148/rg.2016150120. Epub 2016 Feb 12. PMID 26871986
- [Background] Harvey LA, Fornusek C, Bowden JL, Pontifex N, Glinsky J, Middleton JW, Gandevia SC, Davis GM. Electrical stimulation plus progressive resistance training for leg strength in spinal cord injury: a randomized controlled trial. Spinal Cord. 2010 Jul;48(7):570-5. doi: 10.1038/sc.2009.191. Epub 2010 Jan 12. PMID 20065991
- [Background] Kouwijzer I, van der Meer M, Janssen TWJ. Effects of trunk muscle activation on trunk stability, arm power, blood pressure and performance in wheelchair rugby players with a spinal cord injury. J Spinal Cord Med. 2022 Jul;45(4):605-613. doi: 10.1080/10790268.2020.1830249. Epub 2020 Nov 9. PMID 33166206
- [Background] Herzog T, Swanenburg J, Hupp M, Mittaz Hager AG. Effect of indoor wheelchair curling training on trunk control of person with chronic spinal cord injury: a randomised controlled trial. Spinal Cord Ser Cases. 2018 Mar 21;4:26. doi: 10.1038/s41394-018-0057-8. eCollection 2018. PMID 29581893
- [Background] Sliwinski MM, Akselrad G, Alla V, Buan V, Kaemmerlen E. Community exercise programing and its potential influence on quality of life and functional reach for individuals with spinal cord injury. J Spinal Cord Med. 2020 May;43(3):358-363. doi: 10.1080/10790268.2018.1543104. Epub 2018 Nov 26. PMID 30475164
- [Background] Masani K, Sin VW, Vette AH, Thrasher TA, Kawashima N, Morris A, Preuss R, Popovic MR. Postural reactions of the trunk muscles to multi-directional perturbations in sitting. Clin Biomech (Bristol). 2009 Feb;24(2):176-82. doi: 10.1016/j.clinbiomech.2008.12.001. Epub 2009 Jan 18. PMID 19150744
- [Background] McLachlan AJ, McLean AN, Allan DB, Gollee H. Changes in pulmonary function measures following a passive abdominal functional electrical stimulation training program. J Spinal Cord Med. 2013 Mar;36(2):97-103. doi: 10.1179/2045772312Y.0000000031. PMID 23809523